CLINICAL TRIAL: NCT02627950
Title: Impact of Morphine Treatment on Platelet Inhibition in Acute Myocardial Infarction
Acronym: MonAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ingo Eitel, Deputy Director, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-14-10498
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Metoclopramide; Ticagrelor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isotonic sodium chloride + Ticagrelor (Active Comparator): 46 patients with NaCl i.v. and 180 mg ticagrelor orally pre revascularization plus medical standard therapy
  Interventions: Drug: Ticagrelor; Drug: Isotonic sodium chloride
- Morphinhydrochloricum + Ticagrelor (Experimental): 46 patients with 5 mg morphine i.v. and 180 mg ticagrelor pre revascularization plus medical standard therapy
  Interventions: Drug: Morphinhydrochloricum; Drug: Ticagrelor
- Morphinhydrochloricum + Ticagrelor + Metoclopramide (Experimental): 46 patients with 5 mg morphine i.v. and 10 mg MCP i.v. and 180 mg ticagrelor pre revascularization plus medical standard therapy
  Interventions: Drug: Morphinhydrochloricum; Drug: Metoclopramide; Drug: Ticagrelor

INTERVENTIONS:
Drug: Morphinhydrochloricum — 5 mg morphine intravenously
  Other Names: Morphin-hameln (manufacturer: hameln pharmaceuticals)
  Arms: Morphinhydrochloricum + Ticagrelor; Morphinhydrochloricum + Ticagrelor + Metoclopramide
Drug: Metoclopramide — 10 mg MCP intravenously
  Other Names: MCP-ratiopharm (manufacturer: Ratiopharm)
  Arms: Morphinhydrochloricum + Ticagrelor + Metoclopramide
Drug: Ticagrelor — 180 mg ticagrelor orally
  Other Names: Brilique (manufacturer: AstraZeneca)
Drug: Isotonic sodium chloride — 10 ml NaCl 0.9% intravenously
  Other Names: NaCl (manufacturer: Berlin-Chemie Menarini)
  Arms: Isotonic sodium chloride + Ticagrelor

SUMMARY:
The current prospective, randomized, controlled MonAMI trial aims to systematically examine the effects of morphine on the platelet inhibitory effects of the orally administered platelet inhibitor ticagrelor in patients with acute myocardial infarction. In addition, the potential positive or negative effects of MCP in combination with morphine on platelet inhibition will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. ST-elevation myocardial infarction < 24 h after symptom onset or non-ST-elevation myocardial infarction with persistent chest pain < 24 h after symptom onset
2. Intended revascularization by primary percutaneous coronary intervention
3. Informed consent
4. Age ≥18 years

Exclusion Criteria:

1. Age <18 years
2. Active bleeding or bleeding diathesis
3. Oral anticoagulation
4. Current treatment with clopidogrel/prasugrel/ticagrelor/glycoprotein-IIb-IIIa-receptor-antagonists
5. Current treatment with morphine and/or MCP <12 h
6. Contraindication for treatment with platelet inhibitors
7. Fibrinolysis <48 h
8. Percutaneous coronary intervention or coronary artery bypass grafting <3 months
9. Known glomerular filtration rate <30 ml/min
10. Severe liver dysfunction
11. Hypersensitivity to ticagrelor or any excipients
12. History of intracranial hemorrhage
13. Known pregnancy, breast-feeding or intend to become pregnant during the study period
14. Participation in other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Platelet activity 2 hours after administration of loading dose of ticagrelor measured by VerifyNow-P2Y12-test | 2 hours

SECONDARY OUTCOMES:
Platelet reactivity 0.5, 1, 4, 6 and 24 hours after loading dose of ticagrelor measured by VerifyNow-P2Y12-test | 0.5, 1, 4, 6 h and 24 hours
Platelet reactivity 0.5, 1, 2, 4, 6 and 24 hours after loading dose of ticagrelor measured by Vasodilator Stimulated Phosphoprotein-test | 0.5, 1, 2, 4, 6 h and 24 hours
Percentage of patients with high on-treatment platelet reactivity 0.5, 1, 2, 4, 6 and 24 hours after loading dose of ticagrelor (measured by VerifyNow-P2Y12-test) | 0.5, 1, 2, 4, 6 h and 24 hours
Ticagrelor plasma levels and levels of active serum metabolites after 0.5, 1, 2, 4, 6 and 24 hours | 0.5, 1, 2, 4, 6 h and 24 hours
Infarct size measured by delayed enhancement magnetic resonance imaging | Day 1-4
Microvascular obstruction measured by delayed enhancement magnetic resonance imaging | Day 1-4
  Cardiac magnetic resonance imaging equivalent of angiographic no-reflow, expressed as percentage of left ventricular mass

CONTACTS AND LOCATIONS:
Locations (1):
- University of Luebeck, Lübeck, Germany

REFERENCES:
- [Derived] Stiermaier T, Schaefer P, Meyer-Saraei R, Saad M, de Waha-Thiele S, Poss J, Fuernau G, Graf T, Kurz T, Frydrychowicz A, Barkhausen J, Desch S, Thiele H, Eitel I. Impact of Morphine Treatment With and Without Metoclopramide Coadministration on Myocardial and Microvascular Injury in Acute Myocardial Infarction: Insights From the Randomized MonAMI Trial. J Am Heart Assoc. 2021 May 4;10(9):e018881. doi: 10.1161/JAHA.120.018881. Epub 2021 Apr 26. PMID 33899498
- [Derived] Saad M, Meyer-Saraei R, de Waha-Thiele S, Stiermaier T, Graf T, Fuernau G, Langer HF, Kurz T, Poss J, Barkhausen J, Desch S, Eitel I, Thiele H. Impact of Morphine Treatment With and Without Metoclopramide Coadministration on Ticagrelor-Induced Platelet Inhibition in Acute Myocardial Infarction: The Randomized MonAMI Trial. Circulation. 2020 Apr 21;141(16):1354-1356. doi: 10.1161/CIRCULATIONAHA.119.042816. Epub 2020 Apr 20. No abstract available. PMID 32310699